CLINICAL TRIAL: NCT05938296
Title: A Phase 1, Open-label Study of BS006, an Oncolytic Virus, Administered by Intratumoral Injection in Patients With Advanced/Metastatic Solid Tumors
Brief Title: oHSV2-PD-L1/CD3-BsAb Administered Via Intratumoral Injection
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategy adjustment
Sponsor: Binhui Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH-BS006-001
Record Dates: First submitted 2023-06-26; First posted 2023-07-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BS006 injection (Experimental): Subjects will receive BS006 every two weeks, and up to 4mL BS006 will be given. BS006 will be given intratumorally.
  Interventions: Drug: BS006 Injection

INTERVENTIONS:
Drug: BS006 Injection — BS006 will be given every two weeks, and up to 4mL in each treatment. There will be three dose levels: 1×10^6 CCID50/mL, 5×10^6 CCID50/mL, 1×10^7 CCID50/mL.
  Other Names: oHSV2-PD-L1/CD3-BsAb

SUMMARY:
This study will be a Phase 1, multi-center, open-label, dose escalation followed by the recommended phase 2 dose (RP2D) expansion study to characterize safety, tolerability, biodistribution, virus shedding and preliminary efficacy of intratumoral injection of BS006 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Eligible patients are those who have measurable solid tumors as detected by CT or MRI that have persisted, recurred, or metastasized despite therapy. Patients must have histologically confirmed advanced and/or metastatic melanoma, cutaneous squamous cell carcinoma and other solid tumors with palpable, visible or ultrasound detectable lesions. Also, patients with solid tumors that are refractory to standard therapy and for which no existing conventional therapy are eligible. Melanoma patients who were previously treated with IMLYGIC (Talimogene laherparepvec, T-Vec) but did not achieve an optimal response to T-Vec are eligible to receive BS006.

The study will be conducted in 2 parts as described below. Both parts will consist of a screening period of up to 28 days, a treatment period and a follow-up period (safety and long-term follow up). Treatment period of Part 1 will include an initial treatment period (3 doses of BS006) and an optional extended treatment period (repeated every 2 weeks). Subjects will be treated for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 18 years old.
2. Subject must have histologically-only or histologically and cytologically confirmed diagnosis of solid tumors with palpable, visible or ultrasound detectable lesions (e.g., malignant melanoma, cutaneous squamous cell carcinoma and carcinoma of the breast).

   Subjects with tumors that are only confirmed by cytology are not eligible for this trial. Part 2 will only enroll subjects with advanced melanoma or CSCC.
3. Subject must have received and failed all available standard-of-care (SOC) therapies.

   Subjects who are intolerant to treatment with available therapies that are known to confer clinical benefit, or who are intolerant to treatment, or who refuse standard treatment will also be eligible for this study.
4. Subject has measurable disease as determined by RECIST version 1.1. At least 1 lesion must be suitable for intratumoral injection. Lesions for injection must be ≥ 10 mm and ≤ 60 mm in longest diameter.
5. Melanoma patients who were previously treated with IMLYGIC (Talimogene laherparepvec, T-Vec) are eligible after discontinuing the last dose of previous T-Vec treatment for ≥ 12 weeks before first dose of IP.
6. Subjects who have progressed on or are ineligible for available standard therapy are eligible for this trial after the last dose of the previous treatment which is ≥ 4 weeks or 5 half-lives(if required), whichever is longer before the first dose of study treatment.
7. Subject has a predicted life expectancy of ≥ 12 weeks.
8. Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. Men and women of childbearing potential must agree to use adequate contraception from the time of consent through 30 days after final study treatment.Female subject must agree not to breastfeed from screening, throughout the study period and 180 days after the final study drug administration.
10. Females of childbearing potential must have a negative urine or serum pregnancy test within one week prior to start of treatment.
11. Subject must be willing and able to comply with the study requirements including prohibited concomitant medication restrictions.
12. Subject agrees not to participate in another interventional study while receiving study drug.
13. Subject has the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Subject has ongoing toxicity ≥ Common Terminology Criteria for Adverse Events (CTCAE) grade 2 attributable to prior antineoplastic therapies considered clinically significant.
2. Subject has had major surgery ≤ 4 weeks of screening.
3. Subject is concurrently participating in another interventional study or has received an investigational product ≤ 30 days or 5 half-lives prior to first study drug administration.
4. Subject with symptomatic central nervous system (CNS) metastases, except patients with CNS lesions that have been treated and have no evidence of progression in the brain on CT/MRI for ≥ 3 months and have been off steroids for at least 4 weeks prior to first IP administration.
5. Subject with active autoimmune disease requiring systemic therapy within past 2 years (e.g., systemic lupus erythematosus, Wegener syndrome (granulomatosis with polyangiitis),

   Graves' disease, hypophysitis, etc,). The following are exceptions to this criterion:
   * Subject with vitiligo or alopecia
   * Subject with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   * Childhood asthma that has resolved
   * Any chronic skin condition that does not require systemic therapy
   * Type 1 diabetes mellitus ※Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
6. Subject with another malignancy that currently requires treatment.
7. Subject with tumors encasing major vascular structures such as the carotid artery, tumors adjacent to vital neurovascular structures or tumors in locations that are at high risk for AEs or otherwise not considered appropriate for IT injection.
8. Subject with inadequate organ and marrow functions meeting any of the below criteria:

   * Leukocytes < 3000/μL
   * Absolute neutrophil count < 1500/μL (Subjects treated with G-CSF or GM-CSF within 14 days prior to screening will not be enrolled.)
   * Platelets < 100,000/μL (Subjects with a platelet transfusion, or treated with TPO, TPO receptor agonist or IL11 within 14 days prior to screening will not be enrolled.)
   * Hemoglobin (Hgb) < 9 g/dL (Subjects with a blood transfusion or treated with EPO within 14 days prior to screening will not be enrolled.)
   * International normalized ratio (INR) > 1.5 × ULN and/or activated partial thromboplastin time (aPTT) > 1.5 × institutional normal limits
   * Total Bilirubin (TBL) > 1.5 × institutional normal limits (subjects with known Gilbert syndrome who are excluded if TBL > 3.0 × institutional normal limits or direct bilirubin > 1.5 × institutional normal limits)
   * Aspartate aminotransferase (AST) and Alanine transaminase (ALT) > 3.0 × institutional normal limits. Subjects with tumors in the liver AST and ALT > 5 × institutional normal limits.
   * Albumin <3.0 g/dL
   * Estimated glomerular filtration rate (eGFR)<60 mL/min/1.73 m2 (It is calculated according to the CKD-EPI formula)
9. Subject with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of first administration of study drug. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
10. Subject has an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (e.g., subjects with active herpetic skin lesions or prior complications of herpetic infection (e.g., herpetic keratitis or encephalitis), or subjects requiring intermittent or chronic systemic (intravenous or oral) treatment with an anti-herpetic drug (e.g., acyclovir), other than intermittent topical use), symptomatic congestive heart failure, any form of substance abuse or psychiatric illness/social situations that would limit compliance with study visits or requirements, or a condition that could invalidate communication with the Investigator.
11. Subject is known to be positive for human immunodeficiency virus, hepatitis B surface antigen, hepatitis B core immunoglobulin or immunoglobulin G (IgG) antibody, or hepatitis C (IgG or ribonucleic acid (RNA) test) indicating acute or chronic infection.
12. Subject has a history of moderate to severe ascites, clinically significant and/or rapidly accumulating ascites, bleeding esophageal varices, hepatic encephalopathy, or pericardial and/or pleural effusions related to liver insufficiency within 6 months of screening. Mild ascites that does not preclude safe IT injection of BS006 is allowed.
13. Subject has a clinically significant abnormal electrocardiogram (ECG) at screening.
14. Subject has symptomatic cardiovascular disease within the preceding 12 months unless cardiology consultation and clearance has been obtained for study participation, including but not limited to the following: significant coronary artery disease (e.g., requiring angioplasty or stenting), acute myocardial infarction or unstable angina pectoris < 3 months prior to screening, uncontrolled hypertension, clinically significant arrhythmia, or congestive heart failure (New York Heart Association grade ≥ 2).
15. Subject who has a history of bleeding diathesis, are on anti-coagulation therapy, or have abnormal coagulation-fibrinolytic parameters (e.g., activated partial thromboplastin time (APTT), prothrombin time (PT), thrombin time (TT), and platelet count).
16. Subject has medical conditions that predispose the subject to untoward medical risk in the event of volume loading (e.g., intravenous fluid bolus infusion), tachycardia, or hypotension during or following treatment with BS006.
17. Subject has a known or suspected hypersensitivity to BS006 or any components of the formulation used, including prior adverse reaction to vaccinia (e.g., as smallpox vaccine).
18. Subject has had previous exposure with BS006

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2026-12-19 (Estimated); Study Completion 2026-12-19 (Estimated)

PRIMARY OUTCOMES:
Incidence of AE (Adverse Event) and SAE (Serious Adverse Event) | Through study completion, an average of about 1 year(a maximum treatment duration of one year)
  Toxic reactions according to the NCI-CTCAE 5.0 grading standard that occur within 3 weeks from the first administration, are judged to be drug-related by the investigator, and meet the non-hematological toxicity and hematological toxicity conditions specified in the clinical protocol
MTD | up to 1 year
  To estimate the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of BS006

SECONDARY OUTCOMES:
ORR | up to 1 year
  Determination of the ORR is calculated based on the proportion of patients achieving CR or PR using the RECIST v1.1 and modified WHO response criteria as assessed.
DCR | up to 1 year
  DCR is defined as the percentage of participants with a best overall response of CR, PR, or SD.
Biological activity | up to 1 year
  Granulocyte macrophage colony stimulating factor PD-L1/CD3 bispecific antibody mRNA expression in fine needle aspirate (FNA)(Only for Part 1)
Biodistribution | 3 months
  BS006 DNA copy
Viral shedding | 3 months
  BS006 DNA copy

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Orlando Health Cancer Institute, Orlando, Florida
  - Barbara Ann Karmanos Cancer Hospital dba Karmanos Cancer Center, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No